CLINICAL TRIAL: NCT05140005
Title: GlowTest COVID-19 Antigen Home Test Kit Usability Study
Brief Title: GlowTest COVID-19 Antigen Home Test Kit QRI Use Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Arion Bio (Industry)
Collaborators: CSSi Life Sciences (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: AB-001-01
Record Dates: First submitted 2021-11-29; First posted 2021-12-01 (Actual); Last update posted 2021-12-20 (Actual); Status verified 2021-12

CONDITIONS: Covid 19
Keywords: Virus
MeSH Terms: conditions — COVID-19; Virus Diseases

STUDY DESIGN:
Intervention Model Description: 30 subjects split evenly into two sections: 15 participants testing themselves and 15 participants testing another person (child).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- 15 subjects testing themselves (Other): 15 subjects will use the Glow Test Kit to test themselves for Covid 19.
  Interventions: Diagnostic Test: GlowTest COVID-19 Antigen Home Test
- 15 subjects testing someone else (Other): 15 subjects will use the Glow Test Kit to test someone else (a child) for Covid 19.
  Interventions: Diagnostic Test: GlowTest COVID-19 Antigen Home Test

INTERVENTIONS:
Diagnostic Test: GlowTest COVID-19 Antigen Home Test — diagnostic testing for Covid 19
  Other Names: GlowTest

SUMMARY:
The objective of the study is to determine the usability of the GlowTest COVID-19 Antigen Home Test in a simulated home use environment. This is an open label study to evaluate the usability of the GlowTest COVID-19 Antigen Home Test using information from the Quick Reference Instructions and website.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the usability of the GlowTest COVID-19 Antigen Home Test in Home Use. The Arion Bio GlowTest COVID-19 Antigen Home Test is a lateral flow immunoassay intended for the qualitative detection of SARS-CoV-2 nucleocapsid protein antigens from individuals with or without symptoms or other epidemiological reasons to suspect a COVID-19 infection. The test is intended for non-prescription home use with self-collected direct anterior nares swab samples from individuals ages 14 years and older or adult collected anterior nares swab samples from individuals aged 2 to 13. The objective of the study is to determine the usability of the GlowTest COVID-19 Antigen Home Test in a simulated home use environment. This is an open label study to evaluate the usability of the GlowTest COVID-19 Antigen Home Test using information from the Quick Reference Instructions and website.

30 subjects (including both English speaking and Spanish speaking) will be split evenly into two sections: 15 participants testing themselves and 15 participants testing another person (child). There will be one testing site in the United States (US).

ELIGIBILITY:
Inclusion Criteria:

* An Institutional Review Board (IRB) approved informed consent/assent is signed and dated prior to any study-related activities.
* Males and females ages 2 and older.
* Subject is willing to provide a self-collected nasal swab sample. (If under the age of 14, the sample will be collected by an adult.)
* Subject agrees to complete all aspects of the study

Exclusion Criteria:

* Subject has a visual impairment that cannot be restored with glasses or contact lenses.
* Subject has prior medical or laboratory training.
* Subject uses home diagnostics, e.g., glucose meters, HIV tests.
* Subject has prior experience with home COVID test kits.

Min Age: 2 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2021-12-06 (Actual); Primary Completion 2021-12-14 (Actual); Study Completion 2021-12-17 (Actual)

PRIMARY OUTCOMES:
QRI Usability - Observer | 90 minutes
  Assess the usability of the Quick Reference Instructions (QRI) based upon observer evaluation.
QRI Usability - Participant | 90 minutes
  Assess the usability of the kit for home use based upon participant evaluation.

CONTACTS AND LOCATIONS:
Overall Officials: Steven Geller, MD, Principal Investigator — Centennial Medical Group
Locations (1):
- Centennial Medical, Elkridge, Maryland, United States

IPD SHARING:
Plan to Share IPD: No